CLINICAL TRIAL: NCT00655902
Title: Copenhagen Obesity Risk Assessment Study - A Double Blind Randomized Dietary Intervention Study Examining the Effect of a High Intake of Trans Fatty Acids on Abdominal Obesity and Risk Markers of Type 2 Diabetes and Cardiovascular Disease.
Brief Title: Copenhagen Obesity Risk Assessment Study
Acronym: COBRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Dr. med, prof. Arne Astrup, Department of Human Nutrition, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B237
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Metabolic Syndrome; Abdominal Obesity; Heart Disease; Type 2 Diabetes
Keywords: Trans fat; Obesity; Insulin sensitivity
MeSH Terms: conditions — Metabolic Syndrome; Obesity, Abdominal; Heart Diseases; Diabetes Mellitus, Type 2; Obesity; Insulin Resistance | interventions — Trans Fatty Acids; Soybean Oil; Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: Trans fat (soy bean oil)
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Control fat (sunflower oil)

INTERVENTIONS:
Dietary Supplement: Trans fat (soy bean oil) — Industrially produced trans fatty acid from soy bean oil (15 g/d for 16 weeks). The fat (a total of 25 g/d) will be baked into buns.
  Arms: 1
Dietary Supplement: Control fat (sunflower oil) — Control fat from sunflower oil, with 60% oleic acid (in total 25 g/d for 16 weeks). The fat will be baked into buns.
  Arms: 2

SUMMARY:
The aim of the present study is to assess the effect of a high intake of industrially produced trans fatty acids for 16 weeks on abdominal obesity and risk markers of type 2 diabetes and heart disease in healthy, moderately overweight, postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-70 years
* BMI 25-32
* Waist circumference > 80 cm
* Postmenopausal for at least 1 year

Exclusion Criteria:

* BP > 160/100 mmHg
* Fasted blood glucose > 7 mM
* Fasted LDL-cholesterol > 6 mM
* Fasted triglycerides > 3 mM
* Diabetes mellitus or other chronic diseases
* Current or previous cardiovascular disease
* Weight change > 3 kg within last 2 months
* Use of anti-hypertensive drugs
* Use of statins/fibrates
* Use of fish oil supplements
* Smoking
* Hard physical activity > 10 h/week

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
change in LDL-cholesterol/LDL-cholesterol ratio | week 0, 8, 16 and 28
Change in Liver fat measured by MR-S | week 0, 16 and 28
Change in Insulin sensitivity (ISI composite) from 3h OGTT | week 0, 8, 16 and 28

SECONDARY OUTCOMES:
Change in Waist circumference | week 0, 8, 16 and 28
Change in Visceral adipose tissue measured by MR | week 0, 16 and 28
Change in Intramuscular fat measured by MR-S (Psoas Major) | week 0, 16 and 28
Change in Body fat percentage measured by DEXA | week 0, 16 and 28
Change in 24h heart rate variability measured by Holter-monitoring | week 0, 16 and 28
Changes in Cytokines in blood | week 0, 8, 16 and 28
Changes in Cytokines in abdominal adipose tissue | week 0, 16 and 28
Changes in Ceramide in abdominal adipose tissue | week 0, 16 and 28
Changes in Metabolomic profile in blood and urine | week 0, 16 and 28

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Human Nutrition, University of Copenhagen, Frederiksberg, Copenhagen, Denmark

REFERENCES:
- [Result] Bendsen NT, Haugaard SB, Larsen TM, Chabanova E, Stender S, Astrup A. Effect of trans-fatty acid intake on insulin sensitivity and intramuscular lipids--a randomized trial in overweight postmenopausal women. Metabolism. 2011 Jul;60(7):906-13. doi: 10.1016/j.metabol.2011.01.009. Epub 2011 Mar 11. PMID 21397284
- [Result] Bendsen NT, Chabanova E, Thomsen HS, Larsen TM, Newman JW, Stender S, Dyerberg J, Haugaard SB, Astrup A. Effect of trans fatty acid intake on abdominal and liver fat deposition and blood lipids: a randomized trial in overweight postmenopausal women. Nutr Diabetes. 2011 Jan 31;1(1):e4. doi: 10.1038/nutd.2010.4. PMID 23154296
- [Derived] Gurdeniz G, Rago D, Bendsen NT, Savorani F, Astrup A, Dragsted LO. Effect of trans fatty acid intake on LC-MS and NMR plasma profiles. PLoS One. 2013 Jul 29;8(7):e69589. doi: 10.1371/journal.pone.0069589. Print 2013. PMID 23922748
- [Derived] Bendsen NT, Stender S, Szecsi PB, Pedersen SB, Basu S, Hellgren LI, Newman JW, Larsen TM, Haugaard SB, Astrup A. Effect of industrially produced trans fat on markers of systemic inflammation: evidence from a randomized trial in women. J Lipid Res. 2011 Oct;52(10):1821-8. doi: 10.1194/jlr.M014738. Epub 2011 Jul 27. PMID 21795740